CLINICAL TRIAL: NCT05520411
Title: Examining the Effectiveness of Digestive Enzymes at Reducing Bloating and Stomach Distension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HUM Nutrition, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20240
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Stomach Distended; Bloating
Keywords: digestion; bloating
MeSH Terms: conditions — Gastric Dilatation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HUM Flatter Me (Experimental): Come to Citruslabs Office twice (1 Week Gap Between Visits) Visit 1: Take Placebo or Test Product; Eat Test Meal; Outcome Measures Visit 2: Take Placebo or Test Product; Eat Test Meal; Outcome Measures
  Interventions: Dietary Supplement: HUM Flatter Me

INTERVENTIONS:
Dietary Supplement: HUM Flatter Me — Proprietary Enzyme Blend: Protease 3.0 Protease 4.5 Protease 6.0 Neutral Bacterial Protease Peptidase Bromelain Papain Lipase Amylase Glucoamylase Alpha-galactosidase Invertase Diastase Hemicellulase + Cellulase Beta-Glucanase Phytase Lactase Ginger Root Fennel Seed Peppermint Leaf

SUMMARY:
Flatter Me is a product that includes digestive enzymes in a way to support digestion of macronutrients and their constituents and provides herbs traditionally used for digestive health support. This trial aims to test Flatter Me against a placebo pill to examine differences in both subjective outcomes (feelings of bloating and indigestion) and changes in waist circumference (abdominal distension) after eating a test meal.

ELIGIBILITY:
Inclusion Criteria:

* Self Report bloating or stomach distension at least once per day after eating

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Currently taking any prescribed medication meant to treat gut health
* Currently taking any medication for fluid balance (i.e., Aldactone)
* Currently suffers from any pre-existing condition that would prevent them from adhering to the protocol.
* Currently suffers from any pre-existing condition that would prevent them from consuming cheese pizza.
* Use of an antibiotic in the previous 3 months.
* Taking an iron supplement with > 65mg of iron in the last week.
* Diagnosed with any of IBS, chronic constipation, GERD, Crohn's Disease, ulcerative colitis, celiac disease, liver disease, kidney disease, heart failure.
* Lactose Allergy or Intolerance
* Any food allergies
* Current smoker
* Wears dentures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Perceived Changes in Bloating and Stomach Distention | 1 Week
  Questionnaires will be administered to participants at multiple time points before and after eating a test meal. Symptom severity is rated on a scale of 0 (None) to 4 (Extremely Severe)

SECONDARY OUTCOMES:
Visible changes in stomach distension. | 1 week
  Participants will have their waist measured at multiple time points while in the lab

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, PhD, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided